CLINICAL TRIAL: NCT03611842
Title: Study of the Expression of MMPs (Metalloproteinase Matricial) in OME (Otitis Media With Effusion) in Children Under Twelve Years Old With Atrophy of the Eardrum
Brief Title: Study of the Expression of MMPs in OME in Children With Atrophy of the Eardrum
Acronym: MMP and OME
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INM : institut des neurosciences Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0306
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2018-07

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Middle ear effusion fluids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy eardrum: OME (otitis media with effusion)with normal tympanic membrane
  Interventions: Other: preservation of mucosal otitis media
- Atrophic eardrum: OME (otitis media with effusion) with atrophic membrane : thinning of the membrane, retraction pocket
  Interventions: Other: preservation of mucosal otitis media

INTERVENTIONS:
Other: preservation of mucosal otitis media — Suction of the middle ear fluid and conservation of the fluid to be collected instead of thrown away into children Healthy eardrum and Atrophic eardrum

SUMMARY:
Metalloproteinases (MMPs) constitute a family of endopeptidases that cleaves the extracellular matrix as collagen included in the eardrum. Activity of MMP has been shown in some otitis media with effusion (OME) fluids. These enzymes could be directly linked to the prosnostic of OME as it may damage the eardrum and leads to tympanic atrophy.

The main goal of the study is to find out the correlation between activity of MMPs and tympanic atrophy. The investigator will also study if there is any clinical predictive factors in relation to the level of MMPs.

DETAILED DESCRIPTION:
The investigator will include 35 children under 12 years old with OME and who need tympanostomy or tube placement under general anesthesia. Middle ear effusion will be collected, divided in two and frozen.

The investigator will perform ELISA tests to measure the level of MMP2 MMP9 MMP7 et TIMP2 (inhibitor of MMPs). The investigator want to compare the level of MMPs between healthy eardrum and atrophic membrane.

Clinical data will be collected such as age, gender, chronicity of the OME, quality of the eardrum and middle ear effusion type to see if there is any difference when MMPs level is higher.

ELIGIBILITY:
Inclusion Criteria:

- every children under 12 yo operated on in Gui de Chauliac Hospital

Exclusion criteria:

- when effusion is not possible to collect (too thick or amount of fluid not enough)

Collection of both MEE on each ear when OME is bilateral. We will perform the tests on only one ear. The other one will be kept in case of technical issue. A random draw will establish which ear will be tested.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of twelve with OME and surgical indication for myringostomy of tube placement
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Microscopic evaluation of the quality of the eardrum : normal or atrophic | before surgery
  Microscopic evaluation of the quality of the eardrum : normal or atrophic

SECONDARY OUTCOMES:
biochemical assay of the level of TIMP | 1 day
  biochemical assay of the level of TIMP
biochemical assay of the level of MMPs | 1 day
  biochemical assay of the level of MMPs

CONTACTS AND LOCATIONS:
Overall Officials: Lylou Casteil Baume, ENT resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France